CLINICAL TRIAL: NCT03759431
Title: A Randomized Study of Vocal-cord Only vs. Complete Laryngeal Radiotherapy for Early Glottic Cancer
Brief Title: Vocal-cord vs. Complete Laryngeal Radiotherapy for Early Glottic Cancer
Acronym: VOCAL
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: London Health Sciences Centre (Other); M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18.135
Record Dates: First submitted 2018-11-10; First posted 2018-11-30 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Cancer Neck; Larynx Cancer; Glottis Tumor
MeSH Terms: conditions — Head and Neck Neoplasms; Laryngeal Neoplasms

STUDY DESIGN:
Intervention Model Description: Randomized
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Vocal-cord Radiotherapy (Experimental)
  Interventions: Radiation: Vocal-cord Radiotherapy
- Complete Larynx Radiotherapy (Active Comparator)
  Interventions: Radiation: Complete Larynx Radiotherapy

INTERVENTIONS:
Radiation: Vocal-cord Radiotherapy — Focal radiotherapy limited to the involved vocal cord(s) plus additional margins accounting for respiration and set-up errors.
  Arms: Vocal-cord Radiotherapy
Radiation: Complete Larynx Radiotherapy — Radiotherapy to the entire larynx, with target volumes defined to lead to traditional volumes from conventional complete larynx radiotherapy.
  Arms: Complete Larynx Radiotherapy

SUMMARY:
This is a multicentrer, randomized Bayesian Phase II trial for patients with early stage (T1N0) glottic squamous cell carcinoma treated with radical radiotherapy. The primary objective is to assess the non-inferiority of local control achieved with vocal-cord only radiotherapy (VC-RT) compared to complete larynx radiotherapy (CL-RT) in T1N0 glottic laryngeal squamous cell cancer, measured at 2-years after treatment. Secondary outcomes include overall survival, as well as voice impairment, dysphagia and quality of life, measured respectively by the voice handicap index -10 (VHI-10), the MD Anderson Dysphagia Inventory (MDADI) and the MD Anderson Symptom Inventory- Head and Neck module (MDASI-HN). Patients will be randomized in a 1:3 ratio to CL-RT (39 patients) and VC-RT (116 patients) arms. There will be stratification by tumor stage (T1a/T1b) and by institution. An interim analysis is planned after the first 55 patients enrolled on the experimental arm have a 6-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Stage T1a-b N0 of the true vocal cords planned for definitive RT
* Patient not candidate for laser surgery or declined laser surgery
* Biopsy-confirmed squamous cell carcinoma, including verrucous carcinoma
* Eastern Cooperative Oncology Group performance status 0-2
* Ability to provide written informed consent.

Exclusion Criteria:

* Previous irradiation of the head and neck (HNC) region
* Pregnancy or breastfeeding
* Any medical condition that represents, in the opinion of the investigator, a contraindication to radiotherapy or would prevent follow-up after radiotherapy.
* Prior invasive malignancy (except non-melanomatous skin cancer) unless disease free for a minimum of 2 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Estimated)
Dates: Start 2018-10-11 (Actual); Primary Completion 2026-12-12 (Estimated); Study Completion 2026-12-12 (Estimated)

PRIMARY OUTCOMES:
Local control | At 2-year follow-up
  Local control rate of vocal-cord radiotherapy

SECONDARY OUTCOMES:
Voice Handicap Index-10 score | Week 0 post-treatment, and at 2-month, 6-month, 1-year and 2-year follow-up
  Scores are rated on a 0-4 scale to indicate the presence and severity of the symptoms. Lower scores represent better functioning and quality of life.
MD Anderson Dysphagia Inventory score | Week 0 post-treatment, and at 2-month, 6-month, 1-year and 2-year follow-up
  Overall score ranges from 0 to 100, with higher score representing better functioning and quality of life.
MD Anderson Symptom Inventory-Head & Neck score | Week 0 post-treatment, and at 2-month, 6-month, 1-year and 2-year follow-up
  The core and head and neck cancer specific symptoms are rated on a 0-10 scale to indicate the presence and severity of the symptoms. Lower scores represent better functioning and quality of life.
Consensus Auditory-Perceptual Evaluation of Voice (CAPE-V) | Week 0 post-treatment and at 6-month follow-up
  The attributes of CAPE-V are: (a) Overall Severity; (b) Roughness; (c) Breathiness; (d) Strain; (e) Pitch; and (f) Loudness. Each attribute is displayed accompanied by a 100- millimeter line forming a visual analog scale, with a higher score representing more deviant voice attributes.
Rates of acute toxicity as per CTCAE v5.0 | Week 0 post-treatment and at 2-month follow-up
Rates of chronic toxicity as per CTCAE v5.0 | At 6-month, 1-year, 2-year and 5-year post-treatment
Rates of new hypothyroidism | At 2- and 5-year follow-up
Rates of cerebrovascular event (transient ischemic attack or stroke) | At 5-year follow-up
Overall survival | At 2- and 5-year follow-up
Time to recurrence | At 2- and 5-year follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Houda Bahig, Study Chair — Centre hospitalier de l'Université de Montréal (CHUM); David Palma, Study Chair — London Health Sciences Centre
Locations (3):
- The University of Texas MD Anderson Cancer Center, Houston, Texas, United States
- Canada (2):
  - London Health Sciences Centre, London, Ontario
  - Centre Hospitalier de l'Université de Montréal, Montreal, Quebec

REFERENCES:
- [Derived] Bahig H, Rosenthal DI, Nguyen-Tan FP, Fuller DC, Yuan Y, Hutcheson KA, Christopoulos A, Nichols AC, Fung K, Ballivy O, Filion E, Ng SP, Lambert L, Dorth J, Hu KS, Palma D. Vocal-cord Only vs. Complete Laryngeal radiation (VOCAL): a randomized multicentric Bayesian phase II trial. BMC Cancer. 2021 Apr 22;21(1):446. doi: 10.1186/s12885-021-08195-8. PMID 33888069